CLINICAL TRIAL: NCT03161457
Title: A Randomised, Double-blind, Parallel Group, Multicentre Study to Compare the Pharmacokinetics, Pharmacodynamics, Immunogenicity, Safety, and Efficacy of JHL1101 Versus EU-sourced MabThera® in Anti TNF Inadequate Responder Patients With Moderate to Severe Rheumatoid Arthritis (RA) on Background Methotrexate (MTX) Therapy
Brief Title: A Study of JHL1101 Versus MabThera® in Subjects With Severe Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The development was stopped due to company's strategy consideration
Sponsor: JHL Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JHL-CLIN-1101-01
Record Dates: First submitted 2017-04-21; First posted 2017-05-19 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis; Arthritis, Rheumatoid
Keywords: RA; Moderate RA; Moderate Rheumatoid Arthritis; Severe RA; Severe Rheumatoid Arthritis; Moderate to Severe RA; Moderate to Severe Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JHL1101 (Experimental): Each subject will receive 2 intravenous infusions of 1000 mg JHL1101: the first infusion on Baseline and the second on Day 15.
  Interventions: Biological: JHL1101
- MabThera (Active Comparator): Each subject will receive 2 intravenous infusions of 1000 mg MabThera: the first infusion on Baseline and the second on Day 15 (Visit 5).
  Interventions: Biological: MabThera

INTERVENTIONS:
Biological: JHL1101 — 1000 mg containing 10 mg/mL rituximab to be diluted to a concentration of 1 to 4 mg/mL in 0.9% normal saline or 5% D-glucose for administration
  Arms: JHL1101
Biological: MabThera — 1000 mg containing 10 mg/mL rituximab to be diluted to a concentration of 1 to 4 mg/mL in 0.9% normal saline or 5% D-glucose for administration
  Other Names: Rituximab
  Arms: MabThera

SUMMARY:
This is a multicentre, randomised, double-blind, parallel group study to compare the pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, safety, tolerability and efficacy of JHL1101 versus MabThera in subjects with moderate to severe RA who have previously failed at least 1 tumour necrosis factor alpha (TNF) inhibitor (i.e., intolerance or documented active disease despite at least 12 weeks treatment according to the TNF inhibitor-approved treatment and dosage), and are on concomitant treatment with MTX.

DETAILED DESCRIPTION:
This study will take place across approximately 31 centres across 12 countries and will randomise approximately 150 subjects as outpatients.

The primary objective is to investigate and compare the pharmacokinetic profiles of JHL1101 and MabThera (rituximab). The secondary objectives are to investigate the safety, tolerability, and immunogenicity of JHL1101 versus MabThera, to investigate the pharmacodynamics profile of JHL1101 versus MabThera, and investigate the efficacy of JHL1101 versus MabThera.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active RA
* Documented intolerance to or inadequate response to at least 12 weeks of treatment with the licensed regimen of at least one TNF inhibitor therapy
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for at least twelve months after the last dose of study drug.

Exclusion Criteria:

* History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the study drug including known hypersensitivity or allergy to a murine product
* Class IV as per the Classification of Global Functional Status in Rheumatoid Arthritis or wheelchair/bed-bound
* Have any significant systemic involvement with RA such as vasculitis, pulmonary fibrosis or Felty's syndrome
* History of or current inflammatory joint disease other than RA or other systemic disorder where the treatment or current or potential symptoms could confound the assessment of RA, with the exception of secondary Sjögren's syndrome
* Concomitant or recent DMARD treatments for RA
* Oral corticosteroids >10mg/day prednisone equivalent or dose which has not been stable for the 4 weeks prior to Baseline
* Receipt of an intra-articular or other injectable corticosteroid within 4 weeks prior to Screening
* Intolerance or contraindications to IV corticosteroids
* Use of NSAIDs which have not been at a stable dose within 2 weeks prior to Baseline.
* Have undergone surgical treatments for RA including synovectomy and arthroplasty in more than 3 joints and/or within the last 8 weeks prior to Screening
* History of major surgery within the 12 weeks prior to Screening
* History of an infected joint prosthesis which subsequently has not been surgically removed/replaced
* Positive serological test for HBsAg, hepatitis B core antibody or hepatitis C serology.
* History of HIV infection, or a positive test at Screening
* History of tuberculosis (TB) infection.
* Acute clinical manifestations of herpes zoster virus or herpes simplex.
* Active infection of any kind or any major episode of infection requiring hospitalization within 24 week prior to Baseline or requiring treatment with IV anti-infective agents within 8 weeks prior to Baseline or oral anti infective agents within 2 weeks prior to Baseline
* Subjects at risk of progressive multifocal leukoencephalopathy (PML) as per protocol
* Any significant cardiac disease
* Subjects with a history of solid-organ transplantation
* History of lympho- or myeloproliferative disorder or malignancy within the last 5 years

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration versus time curve (AUC) | Day 0 through Week 52
Trough Concentration | Day 15
Maximum Concentration (Cmax) | Day 15

SECONDARY OUTCOMES:
AUC | Up to Week 12
Time to maximum plasma concentration | Day 0 through Week 52
Cmax | Day 0 through Week 52
Total body clearance | Day 0 through Week 52
Volume of distribution | Day 0 through Week 52
Terminal half life | Day 0 through Week 52
Area under plasma concentration versus time curve | Week 2 to Week 24
Incidence of treatment-related adverse events (safety) | Until End-of-Study follow-up at Week 52
Immunogenicity | Baseline, Weeks 12, 16, 24, and 52
  Human anti-chimeric antibody analysis
Area under the depletion-time curve of CD19+ B-cell | Day 0 to Day 15, Day 0 to Week 12, Day 0 to Week 24, and Day 0 to Week 52 (end of study)
Change from Baseline in CD4+ T-cell counts | Day 0 through Week 52
American College of Rheumatology (ACR) criteria 20, 50, 70 response rate | Weeks 4, 8, 12, 16, 24 and 52 and over time from Baseline to Week 52
Swollen and tender joint count | From Baseline to Week 52
Subject's assessment of arthritis pain | From Baseline to Week 52
  2010 ACR/European League Against Rheumatism (EULAR) Classification Criteria for RA

CONTACTS AND LOCATIONS:
Locations (28):
- Bosnia and Herzegovina (2):
  - JHL Biotech Investigational Site, Banja Luka
  - JHL Biotech Investigational Site, Bijeljina
- Bulgaria (2):
  - JHL Biotech Investigational Site, Plovdiv
  - JHL Biotech Investigational Site, Sofia
- JHL Biotech Investigational Site, Prague, Czechia
- Germany (4):
  - JHL Biotech Investigational Site, Bad Doberan
  - JHL Biotech Investigational Site, Hildesheim
  - JHL Biotech Investigational Site, Magdeburg
  - JHL Biotech Investigational Site, Rendsburg
- JHL Biotech Investigational Site, Budapest, Hungary
- JHL Biotech Investigational Site, Vilnius, Lithuania
- Poland (2):
  - JHL Biotech Investigational Site, Poznan
  - JHL Biotech Investigational Site, Wroclaw
- Russia (6):
  - JHL Biotech Investigational Site, Kazan'
  - JHL Biotech Investigational Site, Moscow
  - JHL Biotech Investigational Site, Saint Petersburg
  - JHL Biotech Investigational Site, Samara
  - JHL Biotech Investigational Site, Saratov
  - JHL Biotech Investigational Site, Yaroslavl
- Taiwan (2):
  - JHL Biotech Investigational Site, Taichung
  - JHL Biotech Investigational Site, Taipei
- Ukraine (5):
  - JHL Biotech Investigational Site, Kharkiv
  - JHL Biotech Investigational Site, Kyiv
  - JHL Biotech Investigational Site, Lviv
  - JHL Biotech Investigational Site, Poltava
  - JHL Biotech Investigational Site, Vinnytsia
- United Kingdom (2):
  - JHL Biotech Investigational Site, London
  - JHL Biotech Investigational Site, Southampton